CLINICAL TRIAL: NCT06153108
Title: Monitoring Biomarker for Detecting Change in Physical Activity and Limb Function in Inclusion Body Myositis Over Time
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: BioSensics (Industry)
Responsible Party: Sponsor
Other Study IDs: Biosensics IBM
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Inclusion Body Myositis
Keywords: Biomarker
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PAMSys pendant PAMSys wrist sensors — The PAMSysTM sensor consists of a 3-axis accelerometer, battery, and built-in memory for recording long-term data. Accelerometer data is recorded at a sampling frequency of 50 Hz

SUMMARY:
Inclusion-Body Myositis (IBM) results in weakness and the deterioration of distal arm muscles, the symptoms of which are currently assessed through expert examination at clinical visits. Such in-clinic assessments are time-consuming, subjective, of limited sensitivity, and only provide a snapshot of a patient's disease. In this project, the investigators will conduct clinical validation of monitoring digital biomarkers of upper limb function during activities of daily living using a wearable sensor platform that enables frequent, at-home monitoring of upper limb function health in IBM and could be incorporated into IBM trials.

ELIGIBILITY:
Inclusion Criteria:

1. Meet any of the European Neuromuscular Centre Inclusion Body Myositis research diagnostic criteria 2011 categories for IBM.
2. Able to provide informed consent.

Exclusion Criteria:

1. Unwillingness to follow study procedures.
2. Participation in an investigational drug research study within the past 30 days.

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with diagnosed inclusion body myositis
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Investigate validity of PAMSys wrist sensor and pendant sensor as monitoring biomarker of upper and lower limb function and physical activity, including leg function, change in IBM patients. | Baseline, Month 6, Month 12
  will investigate if sensor-derived parameters measured by the PAMSys wrist sensors and pendant sensor can quantify disease severity and track subtle changes in upper and lower limb health and ambulation over time.

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Dimachkie, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided